CLINICAL TRIAL: NCT00320814
Title: An Exploratory Study of the Safety, Tolerability and Biological Effect of a Single Intravitreal Administration of VEGF Trap in Patients With Diabetic Macular Edema
Brief Title: Phase 1 Study of VEGF Trap in Patients With Diabetic Macular Edema
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Avner Ingerman, MD/Medical Monitor, Regeneron Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGFT-OD-0512
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VEGF Trap-Eye (Experimental): single IVT injection of 4.0 mg of VEGF Trap-Eye into the study eye on Day 1
  Interventions: Drug: VEGF Trap-Eye

INTERVENTIONS:
Drug: VEGF Trap-Eye — single IVT injection of 4.0 mg of VEGF Trap-Eye into the study eye on Day 1

SUMMARY:
To assess the ocular and systemic safety and tolerability of a single intravitreal injection of VEGF Trap in patients with diabetic macular edema.

DETAILED DESCRIPTION:
This is an open label study. Initially, 5 patients with DME will receive an ITV injection of VEGF Trap into the study eye. Additional patients may be enrolled at the same or additional dose levels. Patients will be observed for six weeks following the injection for assessments of ocular and systemic safety.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus (type 1 or type 2).
* Best corrected E-ETDRS visual acuity score of ≥ 24 letters (i.e., 20/320 or better) and ≤ 73 letters (i.e., 20/40 or worse).
* On clinical exam, definite retinal thickening due to diabetic macular edema involving the center of the macula.
* Retinal Thickness at the center point ≥ 250 microns.
* Media clarity, pupillary dilation, and patient cooperation sufficient for adequate fundus photographs.

Exclusion Criteria:

* History of any vitreous hemorrhage within 4 weeks prior to Visit 2 (Day 1).
* Macular edema due to causes other than diabetic macular edema. An eye should be considered ineligible: (1) if the macular edema is considered to be related to cataract extraction or (2) clinical exam and/or OCT suggests that vitreoretinal interface disease (e.g., a taut posterior hyaloid or epiretinal membrane) is the primary cause of the macular edema.
* An ocular condition is present such that, in the opinion of the investigator, visual acuity would not improve from resolution of macular edema (e.g., foveal atrophy, pigmentary changes, dense subfoveal hard exudates, nonretinal condition).
* An ocular condition is present (other than diabetes) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, age-related macular degeneration, uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass Syndrome, etc.).
* Presence of any other condition or laboratory abnormality, which, in the opinion of the Investigator, would interfere with the assessment of disease status/progression or jeopardize the patient's appropriate participation in this Phase 1 study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-04; Primary Completion 2006-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To assess the ocular and systemic safety and tolerability of a single intravitreal (IVT) injection of VEGF Trap-Eye in patients with diabetic macular edema (DME) | Assessments for safety and tolerablity are performed at each visit (Visit 1 - Visit 10)

SECONDARY OUTCOMES:
To obtain a preliminary assessment of the effect of a single dose of VEGF Trap-Eye on central retinal thickness (CRT) at the center point as determined by optical coherence tomography (OCT) | Assessments for CRT are performed at each visit (Visit 1 - Visit 10) by means of OCT.
To obtain a preliminary assessment of the effect of a single IVT administration of VEGF Trap-Eye on visual acuity | Assessments for visual acuity are performed at each visit (Visit 1 - Visit 10).

CONTACTS AND LOCATIONS:
Overall Officials: Avner Ingerman, MD, Study Director — Regeneron Pharmaceuticals
Locations (2):
- United States (2):
  - Baltimore, Maryland
  - Charlotte, North Carolina